CLINICAL TRIAL: NCT05063838
Title: Perioperative Pharmacogenomic Testing (PPGx) : A Feasibility and Randomised Controlled Pilot Study
Brief Title: Perioperative Pharmacogenomic Testing
Acronym: PPGx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: University of Adelaide (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PeterMac ID 20/85
Record Dates: First submitted 2021-09-06; First posted 2021-10-01 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Pharmacogenetics; Anesthesia
Keywords: Drug metabolism; Pharmacogenomics; Individualised care; Postoperative pain; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will remain blinded until the completion of data collection on post-operative day 30. Investigators assessing postoperative outcomes will remain blinded throughout study. Treating clinicians and study investigators will be unblinded to the pharmacogenomic results available for patients randomised to the active arm of the study group. Treating clinicians will remain blinded to the pharmacogenomic results available for patients randomised to the control arm of the study group, as this group will receive standard care that is provided at Peter MacCallum Cancer Centre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacogenomic group (Experimental): The perioperative (anesthetic and postoperative pain management) plan for each patient will be determined preoperatively by the treating anesthesia team. Thereafter, the pharmacogenomic results of the patient will be released and a personalised anesthetic plan formulated based on international pharmacogenomic guidelines. The treating anesthesia team will then modify the perioperative care plan based on the patients' pharmacogenomic results and the international pharmacogenomic guidelines.
  Interventions: Other: Pharmacogenomic optimisation of anaesthetic medications
- Control group (No Intervention): Perioperative care will be managed according to current 'standard care' practice at Peter MacCallum Cancer Centre.

INTERVENTIONS:
Other: Pharmacogenomic optimisation of anaesthetic medications — Personalisation of anaesthetic plan based on pharmacogenomic results and international guidelines.
  Arms: Pharmacogenomic group

SUMMARY:
This is a single centre, prospective feasibility study and pilot randomised controlled trial of patients scheduled for elective intermediate or major non-cardiac surgery. The investigators plan to randomise up to 200 patients who meet the inclusion criteria to standard care or to personalised perioperative care based on pharmacogenomic testing for drugs commonly used in anaesthesia and postoperative pain management e.g., opioids - morphine, oxycodone and tramadol; anti-emetics - metoclopramide and ondansetron; and non-steroidal drugs - celecoxib and ibuprofen.

The investigators hypothesise that pharmacogenomic testing is feasible prior to elective surgery and through 'personalised prescribing' for precision tailored perioperative care the investigators will improve patient's postoperative quality of recovery, including pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Age greater than 18 years
3. Elective surgery scheduled greater than 1 week from preoperative assessment and date of pharmacogenomic testing
4. Moderate-Major surgery expecting to last two or more hours with anticipated admission of at least 1 night including: breast, melanoma, colorectal (laparoscopic or open), prostate, or other major surgery (e.g. oesophagectomy, head and neck cancer, retroperitoneal sarcoma, etc.)

Exclusion Criteria:

1. Day case surgery
2. Expected surgery duration of < 2 hours
3. Urgent surgery expected within 1 week of pre-operative assessment
4. Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - patient acceptability of pre-operative pharmacogenomic testing prior to their scheduled intermediate-major surgery. | Pre-consent
  Percentage of eligible patients approached who consent to participate in the study (yes/no).
Pilot RCT - post-operative pain control on day 1 after surgery | Day 1
  Pain on post-operative day 1 as measured by the Numerical Rating Scale (NRS)

SECONDARY OUTCOMES:
Patient pharmacognemic test result availability prior to surgery (i.e. timely test result availability). | Time of surgery
  Percentage of patient test results available on day of surgery
Patient perceptions of pharmacogenomic testing and reasons patients decline to participate. | Prior to surgery
  Patient questionnaire regarding patient perceptions of pharmacogenomic testing
Actionable genetic variations in our surgical population | Intraoperative
  Frequency of actionable variations as measured by pharmacogenomic testing
Frequency of change of drug prescribing based on pharmacogenomic testing | 72 hours
  Number of changes during the intraoperative period and post-operative period (pharmacogenomic group).
Anesthesia team perceived benefit of modifying perioperative drug choice based on pharmacogenomic results (pharmacogenomic group) | 72 hours
  Percentage of anesthetists who select "I found the pharmacogenomic results helpful in prescribing".
Post-operative pain and nausea and vomiting | 30 days
  Percentage recovery of the nociceptive domain of the PostopQRS™ scale between groups
Quality of recovery during the postoperative period | 30 days
  Percentage recovery over time of all domains of the PostopQRS™.
Quality of recovery on day 1 postoperatively | Day 1
  QoR-15
Post-operative pain as measured by total opioid dose | 72 hours
  Total opioid dose used within the peri-operative period intra-operative, 0-24, 24-48 & 48-72 hours after surgery.
Quality of life at post-operative day 30 | 30 days
  EQ-5D-5L on POD-30 and Days alive at home within 30 days after surgery (DAH-30).

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia